CLINICAL TRIAL: NCT03700931
Title: Episodic Memory Influence on Fruit/Vegetable Consumption in Young Adults With Healthy or Unhealthy Weight
Brief Title: Influence of Episodic Memory on Healthy Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma del Estado de Mexico (Other)
Responsible Party: Principal Investigator, Antonio Laguna Camacho, Full-time Professor, Universidad Autonoma del Estado de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: COFEPRIS 15CI1506014 2018/06
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Eating Behavior
Keywords: Episodic memory; Eating episodes; Fruit and vegetable intake
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: The participants are allocated to one of the two conditions (experimental or control condition) of the study in a randomised sequence.
Who Masked: Participant
Masking Description: The experimental aim is concealed presenting it as a "study on memory of daily activities"
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eating recall condition (Experimental): Participants receive a questionnaire asking them to write down what they ate the day before at breakfast, between breakfasts and lunch, at lunch, between lunch and dinner, at dinner, and after dinner, reporting for each episode the foods and drinks consumed, place, time of the day and people present (10).
  Interventions: Behavioral: Eating recall condition
- Non-eating recall condition (Active Comparator): Participants receive a questionnaire asking them to write down their school, homework (assignment), study, or work-related activities, two at morning, two at afternoon and two at night, of the day before reporting the name of each activity, place, time of the day and people present.
  Interventions: Behavioral: Non-eating recall condition

INTERVENTIONS:
Behavioral: Eating recall condition — Recall of eating episodes would increase subsequent intake of fruit or vegetable items
  Other Names: Cognitive approaches for eating behaviour
  Arms: Eating recall condition
Behavioral: Non-eating recall condition — Recall of non-eating episodes would not influence subsequent intake of fruit or vegetable items
  Arms: Non-eating recall condition

SUMMARY:
The present research project investigates if recall of recent eating episodes enhances consumption of fruits and vegetables

DETAILED DESCRIPTION:
Episodic memory is the capacity to remember past autobiographic events, including eating episodes. Recalling a previous meal decreases the amount eaten in a subsequent snack occasion.

Recall of recent eating episodes could alert individuals about the relationship between their eating behaviour and wellbeing. This is supported by the observation in slimming trials that participants who keep a food diary lose more weight than those who do not record their intake.

Lab experiments have focused on the effect of eating episodic memory on later intake of unhealthy food. However, less is known about the effect on intake of healthy food. Increasing consumption of food that contains nutritious elements like fruit could protect against chronic disease. If eating episodic memory would increase intake of healthy food, this would benefit individuals' health.

The aim of the present between-subjects experiment is to test the influence of memory of recent eating episodes on fruit and vegetable consumption. The interest is to assess differences in amount of fruit/vegetables eaten in each of two conditions: (i) after a recall of eating episodes of the day before and (ii) after recall of activities of the day before excluding eating episodes. The hypothesis is that fruit/vegetable consumption after recalling eating episodes would be higher than after recalling non-eating related activities.

The project will consist of four individual studies varying weight status of participants and test food: i) Female with healthy weight, and fruit as test food; ii) Female with healthy weight, and vegetable as test food; iii) Female with unhealthy weight, and fruit as test food; and iv) Female with unhealthy weight, and vegetable as test food.

ELIGIBILITY:
Inclusion criteria:

* Age 18-25 years old
* Body mass index within ranges of healthy weight and overweight or slight obesity (18.5 to 24.9 and 25.0 to 34.9 kilograms divided by squared height)

Exclusion criteria:

* Fruit hypersensibility
* Vegetable hypersensibility
* Chronic ill health

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Fruit or vegetable intake | One-session intervention, an average of 30 min.
  Amount eaten in grams

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Laguna Camacho, PhD, Principal Investigator — CICMED. Universidad Autónoma del Estado de Mexico
Locations (1):
- Centro de Investigación en Ciencias Médicas, Toluca, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Information about the study is available at the OSF platform
Time Frame: 28 November 2018
URL: https://osf.io/b42te/